CLINICAL TRIAL: NCT00951158
Title: A Molecular Pharmacodynamic Dose-titration Trial of Conjugated Linoleic Acid (CLA; Clarinol®) in Patients With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Administrative suspension. PI/grant holder transferred to new institution.
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D0914; R21CA131820-01A2 (NIH)
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2012-03

CONDITIONS: Advanced Solid Tumors
Keywords: Conjugated Linoleic Acid; Clarinol; S14 Expression
MeSH Terms: interventions — Linoleic Acids, Conjugated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CLA (Experimental): Open-label dose-titration trial of CLA in patients with advanced, refractory malignancies. oral dose 7.5 g/day 28 day cycle
  Interventions: Dietary Supplement: Conjugated Linoleic Acid; Drug: Conjugated Linoleic Acid

INTERVENTIONS:
Dietary Supplement: Conjugated Linoleic Acid — This is a open-label dose-titration trial of CLA in patients with advanced, refractory malignancies. The dose a participant receives is dependent upon the cohort to with the patient is assigned.
  CLA will be given as oral soft gels, once daily, with pharmacokinetic sampling and biopsies (pretreatment and on day 15). Doses will be escalated by patient cohorts, using an accelerated titration design (single-patient cohorts) with expansion to conventional cohort sizes (3-6 patients) once either inhibition of S14 expression or clinical toxicity is observed. Subjects with stable or responsive disease and who tolerate treatment may continue on CLA until the time of disease progression.
  Other Names: CLA; Clarinol
Drug: Conjugated Linoleic Acid — Phase I Dose Escalation Study
  Other Names: Clarinol, CLA

SUMMARY:
It has become apparent that many cancers depend on specific fats (lipids) for their continued growth. Conjugated linoleic acid (CLA) is a safe, popular, and well-tolerated dietary supplement that promotes weight loss and loss of fat. CLA was recently shown to block the metabolism (uptake and production) of lipids required for growth of some cancers, resulting in killing of cancer cells. The investigators will conduct a clinical trial to test whether oral CLA blocks metabolism of lipids in patients with advanced cancers. Since the dose of CLA that may do this is not yet known, the investigators will start at a dose of CLA known to be tolerable and effective for weight loss. If this dose does not block lipid metabolism, the investigators will test higher doses in successive groups of patients until the investigators identify an effective dose, unless the investigators find that these higher doses cannot be tolerated. In order to verify that CLA is absorbed, it is necessary to measure CLA levels in blood before and after doses are given. Likewise, in order to verify that CLA blocks lipid metabolism, the investigators will need to obtain small samples of abdominal fat (and, in some patients, samples of tumors).

ELIGIBILITY:
Inclusion Criteria

A subject is eligible for inclusion in this study only if all of the following criteria apply:

1. Written informed consent.
2. Age 18 years or more.
3. Performance status of 0, 1, or 2 on the Eastern Co-operative Oncology Group (ECOG) Scale.
4. A predicted life expectancy of at least 3 months, in the estimation of the investigator.
5. Subjects with histologically or cytologically confirmed advanced solid tumors, who have failed conventional therapy for their tumor type or have a tumor type for which no standard effective therapy exists.
6. At least 4 weeks since last chemotherapy, radiotherapy, biologic therapy or surgery. Subjects must be free of post-treatment side effects. No concurrent chemotherapy, biologic therapy or radiotherapy is allowed.
7. Hematological/clinical chemistry criteria of:

   Hemoglobin ≥ 9.0 g/dL WBC ≥ 3,500/mm3 [≥ 3.5 x 109/L] Neutrophils ≥ 1,500/mm3 [≥ 1.5 x 109/L] Platelets ≥ 100,000/mm3 [≥ 100.0 x 109/L] Calculated creatinine clearance ≥60 mL/min using the Cockcroft-Gault Formula.
8. Serum bilirubin < 2.0 mg/dL (34 µmol/L)
9. SGOT/AST, SGPT/ALT and alkaline phosphatase < 2 times the upper limit of normal if liver metastases cannot be visualized by abdominal computed tomography (CT) or magnetic resonance imaging (MRI scan). If liver metastases are present, subjects with < 5 times the upper limit of normal are eligible to participate.
10. Once the RP2D is established, additional patients enrolled at the expanded dose cohort must have tumor that is accessible to two serial biopsies and that is documented (by IHC or RT-PCR) to express S14.

Exclusion Criteria

A subject is ineligible if any of the following criteria apply:

1. Cancer cachexia, defined by the combination of: unintentional weight loss ≥10%, low

   caloric intake (≤ 1500 kcal/day), and systemic inflammation (C-reactive protein ≥ 10mg/L).[52]
2. Type II diabetes mellitus
3. Women who are pregnant or lactating, or women subjects of childbearing potential who refuse to practice adequate contraception. (oral contraceptives or IUD; double barrier such as diaphragm plus spermicide; vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner of that female). Childbearing potential is defined as women who are not surgically sterilized (i.e. have not had a hysterectomy, bilateral oophorectomy [ovariectomy], or bilateral tubal ligation) or post-menopausal (i.e., documented absence of menses for one year prior to entry into the study).
4. Men unwilling to abstain from sex or use effective contraception during the study.
5. Subjects with uncontrolled emesis, regardless of etiology.
6. Active infection, or seropositivity for HIV or Hepatitis B/C.
7. Subjects with clinical evidence of any gastrointestinal (GI) conditions (i.e., removal of a portion of the stomach, recent GI obstruction or GI neuropathy) or subjects taking drugs that would alter GI absorption or motility (e.g., cisapride).
8. Intercurrent severe medical problems, which would significantly limit full compliance with the study or expose the subject to unnecessary risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
To define a tolerable dose of oral CLA, given on a daily schedule, that maximally inhibits S14 expression in adipocytes of patients with advanced solid tumors. | 2 years

SECONDARY OUTCOMES:
To quantify the effects of CLA on S14 expression in tumor tissue, at its recommended phase II dose | 2 years
To quantify effects of CLA on expression of lipogenic enzymes regulated by S14, lipoprotein lipase, and phospho-akt in adipocytes (and tumor tissue). | 2 years
To quantify effects of CLA on expression of biomarkers for cellular proliferation, S/G2 phases of cell cycle, and apoptosis in tumor tissue. | 2 years
To define the plasma pharmacokinetics of CLA in patients with advanced cancer. | 2 years
To obtain data on the safety and tolerability of CLA given orally, on a daily schedule to patients with advanced cancer. | 2 years
To document ant tumor activity of CLA, if observed, in this population. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Raymond P Perez, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Norris Cotton Cancer Center, Lebanon, New Hampshire, United States